CLINICAL TRIAL: NCT02079649
Title: A Prospective, Randomized, Double-Masked, Vehicle and Active-Controlled, Safety and Efficacy Study of AL-53817 and AL-78843 Ophthalmic Solutions for the Treatment of Allergic Conjunctivitis in an Environmental Exposure Chamber (EEC) Model
Brief Title: Safety and Efficacy Study of AL-53817 and AL-78843 Ophthalmic Solutions for Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-12-069
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2015-08-06 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic conjunctivitis; Red eyes; Eyelid swelling; Ragweed; Allergies; Itchy eyes; Ocular redness; Chemosis; Tearing; Watery eyes
MeSH Terms: conditions — Conjunctivitis, Allergic; Hypersensitivity; Lacerations | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AL-53817 (Experimental): AL-53817 Ophthalmic Solution, 0.1%, 1 drop in each eye twice daily for 6-8 days followed by 1 drop in each eye once on the last day of dosing (Day 7, 8, or 9)
  Interventions: Drug: AL-53817 Ophthalmic Solution, 0.1%
- AL-78843 (Experimental): AL-78843 Ophthalmic Solution, 0.03%, 1 drop in each eye twice daily for 6-8 days followed by 1 drop in each eye once on the last day of dosing (Day 7, 8, or 9)
  Interventions: Drug: AL-78843 Ophthalmic Solution, 0.03%
- Maxidex (Active Comparator): Dexamethasone Ophthalmic Suspension, 0.1%, 1 drop in each eye twice daily for 6-8 days followed by 1 drop in each eye once on the last day of dosing (Day 7, 8, or 9)
  Interventions: Drug: Dexamethasone Ophthalmic Suspension, 0.1%
- Vehicle (Placebo Comparator): AL-53817 Vehicle, 1 drop in each eye twice daily for 6-8 days followed by 1 drop in each eye once on the last day of dosing (Day 7, 8, or 9)
  Interventions: Drug: AL-53817 Vehicle

INTERVENTIONS:
Drug: AL-53817 Ophthalmic Solution, 0.1%
  Arms: AL-53817
Drug: AL-78843 Ophthalmic Solution, 0.03%
  Arms: AL-78843
Drug: Dexamethasone Ophthalmic Suspension, 0.1%
  Other Names: Maxidex®
  Arms: Maxidex
Drug: AL-53817 Vehicle — Inactive ingredients used for masking purposes
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate two investigational ophthalmic solutions for reduction in ocular redness in subjects with allergic conjunctivitis.

DETAILED DESCRIPTION:
Eligible subjects attended 8 study visits, 5 of which included a 3-hour period of ragweed exposure in an Environmental Exposure Chamber. At the sixth visit, subjects received study product and began dosing for up to 9 days. The final visit was the final day of dosing. Participation in this study lasted up to 68 days.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent
* Use of condom by sexually active males for the entire duration of the study.
* Best corrected visual acuity of 55 or greater in each eye as measured by ETDRS (letters read method).
* Able and willing to comply with study protocol and follow protocol instructions.
* Able to avoid any of the topical ocular or systemic excluded medications during the entire study period.
* At least 1 year subject-reported or physician-diagnosed history (prior to Screen Visit) of allergic conjunctivitis during the ragweed season.
* Positive skin prick test for short ragweed allergen within 12 months prior to Screen Visit.
* Significant staff-assessed ocular redness in at least one region in each eye within the 3 hour period of allergen exposure in the EEC (Screen Visits).
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 1 week following the last dose of investigational product.
* Presence of any ocular infection, history of ocular Herpes (simplex or zoster) or adenoviral infection in either eye.
* History of any ocular infection, physician or subject diagnosed, within 30 days prior to Screen Visit.
* Presence of glaucoma, past history of, or diagnosis of glaucoma or ocular hypertension.
* Presence of blepharitis, active rosacea affecting the ocular adnexa, meibomian gland dysfunction, follicular conjunctivitis, intraocular inflammation, or preauricular lymphadenopathy or any other ophthalmic abnormality that may affect the study outcomes.
* Corneal conditions affecting the corneal structure.
* Unwilling to discontinue contact lens wear during the study period.
* Any ocular surgery including ocular laser procedures within 1 year prior to Screen Visit.
* Current or recent (<6 months prior to Screen Visit) history of severe, unstable, or uncontrolled autoimmune, neurological, cardiovascular, hematological, hepatic, renal, psychological, respiratory, gastrointestinal and/or immunological disease or evidence of other diseases based upon a review of medical history and/or physical examination that, in the opinion of the Investigator, would preclude safe subject participation in the study.
* Receiving treatment for anxiety and/or depression at the Screen Visit; any history of suicide attempt.
* Participation in any investigational study within 30 days of Screen Visit or concomitantly with this study.
* Known contraindications or hypersensitivities to any of the study medications or their components
* Confirmed (by physician or optometrist) diagnosis of dry eye.
* History of sensitivity or adverse reaction to steroids.
* Known allergic reaction that is unresponsive to corticosteroids or non-steroidal anti-inflammatory drugs (NSAIDS).
* Physician diagnosed asthma (except inactive childhood asthma and exercise-induced asthma).
* Evidence of active inflammation in the eye as determined by the dilated fundus examination conducted at Screen C Visit.
* Any corneal swelling or haze as determined by the slitlamp examination conducted at Screen C Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Manager, Pharma, GCRA, Study Director — Alcon Research

REFERENCES:
- [Derived] Jacobs RL, Ramirez DA, Rather CG, Andrews CP, Jupiter DC, Trujillo F, Shulman DG. Redness response phenotypes of allergic conjunctivitis in an allergen challenge chamber. Ann Allergy Asthma Immunol. 2017 Jan;118(1):86-93.e2. doi: 10.1016/j.anai.2016.10.023. PMID 28007090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in the US.
Pre-assignment Details: Of the 224 enrolled, 60 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects. Note: 2 randomized subjects were exited prior to treatment.
Groups:
- AL-78843; AL-53817; Maxidex; Vehicle: One drop in each eye twice daily for 6-8 days followed by 1 drop in each eye once on the last day of dosing (Day 7, 8, or 9)
Period: Overall Study
Arm/Group | AL-78843 | AL-53817 | Maxidex | Vehicle
Started | 42 | 41 | 41 | 40
Treated | 41 | 41 | 40 | 40
Completed | 41 | 41 | 40 | 38
Not Completed | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Randomization error (prior to treatment) | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were randomized to and treated with investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-78843 | AL-53817 | Maxidex | Vehicle | Total
Number analyzed (Participants) | 41 | 41 | 40 | 40 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (13.4) | 46.4 (13.3) | 40.9 (13.1) | 46.0 (12.6) | 44.0 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 24 | 24 | 88
  Male | 20 | 22 | 16 | 16 | 74

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Ocular Redness, Area Under the Curve From Time Zero to Hour 10 [AUC (0-10)] at Day 7
Description: Ocular redness ratings were collected for nasal and temporal areas of each eye and assessed by investigational center staff using a visual scale (ie, scored by comparing the subject's eye with a series of photographs) and graded on a scale from 0 (none) to 4 (extremely severe), 0.5 unit steps permitted. AUC was calculated using the trapezoidal rule with unequal intervals as determined by the assessment time points. Change was calculated as AUC(0-10)[Day 7] - AUC(0-10) [Baseline]. Both eyes contributed to the analysis.
Time Frame: 0.0, 0.25, 0.50, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 7.0, 8.0, 9.0, and 10.0 hours on Days 1 (baseline) and 7
Population: This analysis population includes all randomized subjects who had a baseline evaluation minus those who had important protocol deviations that could have affected the outcome of the study.
Measure: Mean (Standard Error); unit: hours x units on a scale
Arm/Group | AL-78843 | AL-53817 | Maxidex | Vehicle
Number analyzed (Participants) | 41 | 41 | 40 | 38
hours x units on a scale | -2.8 (0.68) | -4.7 (0.68) | -8.1 (0.69) | -4.5 (0.70)

2. Secondary Outcome: Mean Change From Baseline in Ocular Itching, Area Under the Curve From Time Zero to Hour 10 [AUC (0-10)] at Day 7
Description: Ocular itching was assessed by the subject with both eyes rated together and scored on a scale from 0 (none) to 4 (incapacitating itch with irresistible urge to rub). AUC was calculated using the trapezoidal rule with unequal intervals as determined by the assessment time points. Change was calculated as AUC(0-10)[Day 7] - AUC(0-10) [Baseline].
Time Frame: 0.0, 0.25, 0.50, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 7.0, 8.0, 9.0, and 10.0 hours on Days 1 (baseline) and 7
Population: as for outcome 1
Measure: Mean (Standard Error); unit: hours x units on a scale
Arm/Group | AL-78843 | AL-53817 | Maxidex | Vehicle
Number analyzed (Participants) | 41 | 41 | 40 | 38
hours x units on a scale | -7.8 (1.00) | -8.8 (1.00) | -10.7 (1.01) | -8.5 (1.04)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (April 2014 - July 2014). All AEs were obtained as solicited comments from the study subjects and as observations by the study Investigator.
Description: An AE was considered to be any untoward medical occurrence in a subject who was exposed to investigational product or that occurred at any time prior to administration of the first dose of the study treatment. AEs are reported as pre-treatment and treatment-emergent.
Groups:
- Pre-Treatment: Includes all subjects who consented to participate in the study
- AL-78843; AL-53817; Maxidex; Vehicle: Includes all subjects who were randomized to and treated with investigational product
Arm/Group | Pre-Treatment | AL-78843 | AL-53817 | Maxidex | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/41 | 0/41 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/224 | 0/41 | 0/41 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.